CLINICAL TRIAL: NCT04246177
Title: A Phase 3 Multicenter, Randomized, Double-blinded, Active-controlled, Clinical Study to Evaluate the Safety and Efficacy of Lenvatinib (E7080/MK-7902) With Pembrolizumab (MK-3475) in Combination With Transarterial Chemoembolization (TACE) Versus TACE in Participants With Incurable/Non-metastatic Hepatocellular Carcinoma (LEAP-012)
Brief Title: Safety and Efficacy of Lenvatinib (E7080/MK-7902) With Pembrolizumab (MK-3475) in Combination With Transarterial Chemoembolization (TACE) in Participants With Incurable/Non-metastatic Hepatocellular Carcinoma (MK-7902-012/E7080-G000-318/LEAP-012)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7902-012; MK-7902-012 (Other: MSD Protocol Number); LEAP-012 (Other: MSD); E7080-G000-318 (Other: Eisai Protocol Number); 205286 (Registry Identifier: JAPIC-CTI); 2022-502116-36-00 (Registry Identifier: EU CT); U1111-1283-3439 (Registry Identifier: UTN); 2019-002345-37 (EudraCT Number)
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: receptor tyrosine kinase inhibitor; programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lenvatinib plus Pembrolizumab plus TACE (Experimental): Participants will receive a combination of lenvatinib, pembrolizumab, and TACE. Lenvatinib will be administered at a dose of 12 mg (for participants with screening body weight ≥60 kg) or 8 mg (for participants with screening body weight <60 kg) orally once a day during each 21-day cycle until progressive disease or unacceptable toxicity (up to 2 years [~35 cycles] or longer with Sponsor approval). Pembrolizumab will be administered via IV infusion at a dose of 400 mg once every 6 weeks (Q6W) for up to 2 years (~17 doses). Participants will undergo TACE as a background procedure of chemotherapeutic and embolic agent(s).
  Interventions: Drug: Lenvatinib; Biological: Pembrolizumab; Procedure: TACE
- Oral Placebo plus IV Placebo plus TACE (Active Comparator): Participants will receive a combination of lenvatinib-matching oral placebo, pembrolizumab-matching IV placebo, and TACE. Lenvatinib-matching oral placebo will be administered once a day during each 21-day cycle for up to 2 years (~35 cycles) or longer with Sponsor approval and pembrolizumab-matching IV placebo will be administered once every 6 weeks (Q6W) for up to 2 years (~17 doses). Participants will undergo TACE as a background procedure of chemotherapeutic and embolic agent(s).
  Interventions: Drug: Oral Placebo; Drug: IV Placebo; Procedure: TACE

INTERVENTIONS:
Drug: Lenvatinib — Administered at a dose of 12 mg (for participants with screening body weight ≥60 kg) or 8 mg (for participants with screening body weight <60 kg) via oral capsules once a day during each 21-day cycle.
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Lenvatinib plus Pembrolizumab plus TACE
Biological: Pembrolizumab — Administered via IV infusion at a dose of 400 mg once every 6 weeks (Q6W).
  Other Names: MK-3475; KEYTRUDA®
  Arms: Lenvatinib plus Pembrolizumab plus TACE
Drug: Oral Placebo — Lenvatinib-matching placebo administered via oral capsules once a day during each 21-day cycle.
  Arms: Oral Placebo plus IV Placebo plus TACE
Drug: IV Placebo — Pembrolizumab-matching placebo administered via IV infusion once every 6 weeks (Q6W).
  Arms: Oral Placebo plus IV Placebo plus TACE
Procedure: TACE — Conducted as a background procedure of chemotherapeutic and embolic agent(s).

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of lenvatinib and pembrolizumab in combination with TACE versus TACE plus oral and intravenous (IV) placebos in participants with incurable, non-metastatic hepatocellular carcinoma (HCC). The primary hypotheses are that pembrolizumab plus lenvatinib in combination with TACE is superior to placebo plus TACE with respect to progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of HCC confirmed by radiology, histology, or cytology
* Has HCC localized to the liver and not amenable to curative treatment
* Participants with Hepatitis C virus (HCV) are eligible if treatment was completed at least 1 month prior to starting study intervention
* Participants with Hepatitis B virus (HBV) are eligible
* Has adequately controlled blood pressure with or without antihypertensive medications
* Has adequate organ function

Exclusion Criteria:

* Is currently a candidate for liver transplantation
* Has had gastric bleeding within the last 6 months
* Has ascites that is not controlled with medication
* Has significant cardiovascular impairment within 12 months of the first dose of study intervention such as congestive heart failure
* Has a serious nonhealing wound, ulcer, or bone fracture
* Has received locoregional therapy to existing liver lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to ~43 months
  PFS is defined as the time from randomization to the first documented progressive disease or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1 as assessed by blinded independent central review (BICR).
Overall Survival (OS) | Up to ~95 months
  OS is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
PFS per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) | Up to ~43 months
  PFS is defined as the time from randomization to the first documented progressive disease or death due to any cause, whichever occurs first. Responses are according to mRECIST as assessed by BICR.
Objective Response Rate (ORR) per mRECIST | Up to ~95 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of any intratumoral arterial enhancement in all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of viable [enhancement in the arterial phase] target lesions, taking as reference the baseline sum of the diameters of target lesions). Responses are according to mRECIST as assessed by BICR.
Disease Control Rate (DCR) per mRECIST | Up to ~95 months
  DCR is defined as the percentage of participants who have a best overall response of CR (disappearance of any intratumoral arterial enhancement in all target lesions), PR (at least a 30% decrease in the sum of diameters of viable [enhancement in the arterial phase] target lesions, taking as reference the baseline sum of the diameters of target lesions), or stable disease (SD). Responses are according to mRECIST as assessed by BICR.
Duration of Response (DOR) per mRECIST | Up to ~95 months
  DOR is determined by disease assessment and is defined as the time from the first documented evidence of a response of CR (disappearance of any intratumoral arterial enhancement in all target lesions) or PR (at least a 30% decrease in the sum of diameters of viable [enhancement in the arterial phase] target lesions, taking as reference the baseline sum of the diameters of target lesions) until the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to mRECIST as assessed by BICR.
Time to Progression (TTP) per mRECIST | Up to ~95 months
  TTP is defined as the time from randomization to the first documented disease progression. Responses are according to mRECIST as assessed by BICR.
Percentage of Participants Who Experience At Least One Adverse Event (AE) | Up to ~95 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience at least one AE will be reported.
Percentage of Participants Who Experience At Least One Serious Adverse Event (SAE) | Up to ~95 months
  An SAE is an AE that results in death, is life threatening, requires or prolongs a hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, is a cancer, is associated with an overdose, or is another important medical event. The percentage of participants who experience at least one SAE will be reported.
Percentage of Participants Who Experience At Least One Hepatic Event of Clinical Interest (ECI) | Up to ~95 months
  Percentage of participants with Hepatic ECIs not due to disease progression or TACE as assessed by the investigator will be reported.
Percentage of Participants Who Discontinue Study Drug Due to an AE | Up to ~95 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study drug due to an AE will be reported.
ORR per RESCIST 1.1 | Up to ~95 months
  ORR is defined as the percentage of participants who have a confirmed complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by BICR.
DCR per RECIST 1.1 | Up to ~95 months
  DCR is defined as the percentage of participants who have a best overall response of CR (disappearance of all target lesions), PR (at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters), or SD. Responses are according to RECIST 1.1 as assessed by BICR.
DOR per RECIST 1.1 | Up to ~95 months
  DOR is determined by disease assessment and is defined as the time from the first documented evidence of a response of CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters) until the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1 as assessed by BICR.
TTP per RECIST 1.1 | Up to ~95 months
  TTP is defined as the time from randomization to the first documented disease progression. Responses are according to RECIST 1.1 as assessed by BICR.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (205):
- United States (27):
  - Arizona Oncology Associates PC- HOPE ( Site 0770), Tucson, Arizona
  - Scripps Clinic Torrey Pines ( Site 0714), La Jolla, California
  - USC Norris Comprehensive Cancer Center ( Site 0717), Los Angeles, California
  - UCLA Hematology/Oncology - Santa Monica ( Site 0720), Los Angeles, California
  - UC Irvine Health ( Site 0718), Orange, California
  - Yale Cancer Center ( Site 0724), New Haven, Connecticut
  - Tampa General Hospital ( Site 0764), Tampa, Florida
  - Mountain States Tumor Institute ( Site 0773), Boise, Idaho
  - University of Iowa Hospital and Clinics ( Site 0729), Iowa City, Iowa
  - University of Kansas Cancer Center ( Site 0731), Westwood, Kansas
  - University of Louisville ( Site 0757), Louisville, Kentucky
  - Tulane Medical Center ( Site 0787), New Orleans, Louisiana
  - University Medical Center New Orleans ( Site 0733), New Orleans, Louisiana
  - Henry Ford Hospital-GI/Hepatology Research ( Site 0735), Detroit, Michigan
  - Saint Louis University ( Site 0769), St Louis, Missouri
  - University of New Mexico Comprehensive Cancer Center ( Site 0805), Albuquerque, New Mexico
  - Monter Cancer Center ( Site 0780), Lake Success, New York
  - Icahn School of Medicine at Mount Sinai ( Site 0744), New York, New York
  - Wake Forest Baptist Health ( Site 0741), Winston-Salem, North Carolina
  - University of Cincinnati Medical Center ( Site 0791), Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center ( Site 0759), Columbus, Ohio
  - ProMedica Flower Hospital ( Site 0796), Sylvania, Ohio
  - Stephenson Cancer Center ( Site 0745), Oklahoma City, Oklahoma
  - OHSU Center for Health & Healing ( Site 0746), Portland, Oregon
  - Penn State Hershey Medical Center ( Site 0766), Hershey, Pennsylvania
  - Houston Methodist Research Institute ( Site 0784), Houston, Texas
  - Edwards Comprehensive Cancer Center ( Site 0786), Huntington, West Virginia
- Australia (6):
  - St George Hospital ( Site 0005), Kogarah, New South Wales
  - Westmead Hospital-Gastroenterology & Hepatology ( Site 0009), Westmead, New South Wales
  - Princess Alexandra Hospital ( Site 0006), Brisbane, Queensland
  - Austin Health ( Site 0008), Heidelberg, Victoria
  - Alfred Health ( Site 0004), Melbourne, Victoria
  - Royal Perth Hospital ( Site 0002), Perth, Western Australia
- Brazil (8):
  - Liga Norte Riograndense Contra o Câncer-Centro de Pesquisa Clínica ( Site 0057), Natal, Rio Grande do Norte
  - Hospital Nossa Senhora da Conceição-Centro Integrado de Pesquisa em Oncologia ( Site 0056), Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia Reichow ( Site 0052), Blumenau, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos-Unidade de Pesquisa Clínica ( Site 0058), Barretos, São Paulo
  - Fundacao Dr Amaral Carvalho ( Site 0050), Jaú, São Paulo
  - Hospital de Base de Sao Jose de Rio Preto ( Site 0043), São José do Rio Preto, São Paulo
  - BP - A Beneficencia Portuguesa de São Paulo ( Site 0046), São Paulo, São Paulo
  - A.C. Camargo Cancer Center ( Site 0054), São Paulo
- Chile (4):
  - Centro de Oncología de Precisión-Oncology ( Site 0068), Santiago, Region M. de Santiago
  - Centro de Cancer Nuestra Senora de la Esperanza ( Site 0065), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0066), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 0064), Temuco, Región de la Araucanía
- China (39):
  - Anhui Provincial Hospital ( Site 0092), Heifei, Anhui
  - Beijing Cancer Hospital ( Site 0099), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 0105), Beijing, Beijing Municipality
  - Peking Union Medical College Hospital ( Site 0087), Beijing, Beijing Municipality
  - Chinese People s Liberation Army Army Characteristic Medical Center ( Site 0117), Chongqing, Chongqing Municipality
  - Chongqing University Three Gorges Hospital ( Site 0859), Chongqing, Chongqing Municipality
  - Mengchao Hepatobiliary Hospital of Fujian Medical University ( Site 0121), Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital ( Site 0085), Fuzhou, Fujian
  - The First Affiliated Hospital of Fujian Medical University ( Site 0089), Fuzhou, Fujian
  - Zhongshan Hospital Fudan University (Xiamen Branch) ( Site 0133), Xiamen, Fujian
  - Zhujiang Hospital of Southern Medical University ( Site 0115), Guangzhou, Guangdong
  - Guangdong Provincial People s Hospital ( Site 0100), Guangzhou, Guangdong
  - NANFANG HOSPITAL SOUTHERN MEDICAL UNIVERSITY ( Site 0088), Guangzhou, Guangdong
  - SUN YAT-SEN UNIVERSITY CANCER CENTRE ( Site 0128), Guangzhou, Guangdong
  - Jinan University - Zhuhai People's Hospital-Intervention Department ( Site 0856), Zhuhai, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital-Hepatological surgery ( Site 0862), Nanning, Guangxi
  - Hainan General Hospital ( Site 0112), Haikou, Hainan
  - Harbin Medical University Cancer Hospital ( Site 0090), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 0114), Zhengzhou, Henan
  - Tongji Hospital Tongji Medical,Science & Technology ( Site 0126), Wuhan, Hubei
  - Hubei Cancer Hospital ( Site 0101), Wuhan, Hubei
  - Hunan Provincial People's Hospital ( Site 0113), Changsha, Hunan
  - Hunan Cancer Hospital ( Site 0096), Changsha, Hunan
  - The First Affiliated Hospital of Soochow University ( Site 0120), Suzhou, Jiangsu
  - Jiangxi Provincial Cancer Hospital-Cancer Hospital ( Site 0134), Nanchang, Jiangxi
  - Xi'an International Medical Center Hospital ( Site 0860), Xi'an, Shaanxi
  - The Third Affiliated Hospital of the PLA Navy Medical University ( Site 0123), Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center ( Site 0106), Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University ( Site 0084), Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Xi an Jiaotong University ( Site 0108), Xi’an, Shanxi
  - West China Hospital of Sichuan University ( Site 0119), Chengdu, Sichuan
  - Suining Central Hospital ( Site 0857), Suining, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital ( Site 0098), Tianjin, Tianjin Municipality
  - Tianjin Third Central Hospital ( Site 0861), Tianjin, Tianjin Municipality
  - The First Hospital of Kunming ( Site 0124), Kunming, Yunnan
  - 2nd Affil Hosp of Zhejiang University College of Medicine ( Site 0110), Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ( Site 0094), Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital ( Site 0103), Hangzhou, Zhejiang
  - Ningbo Medical Center LiHuili Hospital ( Site 0132), Ningbo, Zhejiang
- Colombia (4):
  - Hospital Pablo Tobon Uribe ( Site 0145), Medellín, Antioquia
  - Administradora Country S.A. ( Site 0137), Bogotá, Bogota D.C.
  - Fundacion Cardiovascular de Colombia ( Site 0136), Piedecuesta, Santander Department
  - Fundación Valle del Lili ( Site 0140), Cali, Valle del Cauca Department
- Denmark (3):
  - Herlev Hospital ( Site 0170), Herlev, Capital Region
  - Aarhus Universitets hospital ( Site 0175), Aarhus N, Central Jutland
  - Odense Universitetshospital ( Site 0160), Odense, Region Syddanmark
- France (6):
  - Hopital de la Croix-Rousse ( Site 0193), Lyon, Auvergne
  - Hopital de la Timone ( Site 0188), Marseille, Bouches-du-Rhone
  - CHU Bordeaux Haut-Leveque ( Site 0185), Pessac, Gironde
  - C.H.U. de Nancy. Hopital de Brabois Adultes ( Site 0180), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - A.P.H. Paris, Hopital Henri Mondor ( Site 0179), Créteil, Val-de-Marne
  - Hopital Paul Brousse ( Site 0182), Villejuif, Val-de-Marne
- Germany (9):
  - Universitaetsklinikum Freiburg ( Site 0199), Freiburg im Breisgau, Baden-Wurttemberg
  - Krankenhaus Nord-West GmbH ( Site 0208), Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover ( Site 0200), Hanover, Lower Saxony
  - Universitaetsklinikum Bonn ( Site 0203), Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Leipzig ( Site 0202), Leipzig, Saxony
  - Universitaetsklinikum Halle ( Site 0213), Halle, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein-Campus Lubeck ( Site 0215), Lübeck, Schleswig-Holstein
  - Charite - Universitaetsmedizin ( Site 0204), Berlin
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0207), Hamburg
- Prince of Wales Hospital ( Site 0242), Shatin, Hong Kong
- Hungary (3):
  - Somogy Megyei Kaposi Mór Oktató Kórház-Oncology center ( Site 0267), Kaposvár, Somogy County
  - Zala Megyei Szent Rafael Korhaz ( Site 0265), Zalaegerszeg, Zala County
  - Semmelweis University ( Site 0264), Budapest
- St Vincents University Hospital ( Site 0690), Dublin, Ireland
- Israel (5):
  - Emek Medical Center ( Site 0307), Afula
  - Rambam Health Care Campus-Oncology Division ( Site 0305), Haifa
  - Hadassah Ein Karem Jerusalem ( Site 0303), Jerusaelm
  - Rabin Medical Center ( Site 0304), Petah Tikva
  - Sourasky Medical Center ( Site 0306), Tel Aviv
- Italy (9):
  - Ospedale del Mare ( Site 0327), Napoli, Campania
  - ASST Grande Ospedale Metropolitano Niguarda-Oncologia Falck ( Site 0331), Milan, Milano
  - Ospedale Mauriziano-SCDU ONCOLOGIA MEDICA ( Site 0333), Turin, Piedmont
  - AOU Policlinico G. Martino ( Site 0324), Messina, Sicily
  - Azienda Ospedaliera Spedali Civili di Brescia-Oncology ( Site 0334), Brescia
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico ( Site 0325), Milan
  - Az Osp di Rilievo Nazionale A. Cardarelli ( Site 0329), Napoli
  - Azienda USL della Romagna-Dipartimento di Oncologia ed Ematologia ( Site 0332), Ravenna
  - Policlinico Universitario -Agostino Gemelli ( Site 0328), Roma
- Japan (25):
  - National Cancer Center Hospital East ( Site 0347), Kashiwa, Chiba
  - Ehime University Hospital ( Site 0368), Tōon, Ehime
  - Kurume University Hospital ( Site 0362), Kurume, Fukuoka
  - Sapporo Kosei General Hospital ( Site 0345), Sapporo, Hokkaido
  - Kanazawa University Hospital ( Site 0354), Kanazawa, Ishikawa-ken
  - Kagawa Prefectural Central Hospital ( Site 0364), Takamatsu, Kagawa-ken
  - Toranomon Hospital Kajigaya ( Site 0369), Kawasaki, Kanagawa
  - Yokohama City University Medical Center ( Site 0351), Yokohama, Kanagawa
  - Kanagawa Cancer Center ( Site 0352), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 0359), Kashihara, Nara
  - Kindai University Hospital ( Site 0358), Sayama, Osaka
  - Saitama Medical University Hospital ( Site 0370), Iruma-gun, Saitama
  - Shizuoka Cancer Center ( Site 0365), Suntogun, Shizuoka
  - Jichi Medical University Hospital ( Site 0353), Shimotsuke, Tochigi
  - Chiba University Hospital ( Site 0346), Chiba
  - National Hospital Organization Kyushu Medical Center ( Site 0361), Fukuoka
  - Hiroshima University Hospital ( Site 0360), Hiroshima
  - Kumamoto University Hospital ( Site 0372), Kumamoto
  - University Hospital,Kyoto Prefectural University of Medicine ( Site 0367), Kyoto
  - Osaka International Cancer Institute ( Site 0357), Osaka
  - Japanese Red Cross Osaka Hospital ( Site 0356), Osaka
  - Saga-Ken Medical Centre Koseikan ( Site 0363), Saga
  - Toranomon Hospital ( Site 0349), Tokyo
  - Juntendo University Hospital ( Site 0371), Tokyo
  - The University of Tokyo Hospital ( Site 0348), Tokyo
- Netherlands (5):
  - Maastricht University Medical Centre ( Site 0440), Maastricht, Limburg
  - AMC ( Site 0438), Amsterdam, North Holland
  - Leids Universitair Medisch Centrum-Medical Oncology ( Site 0442), Leiden, South Holland
  - Erasmus University Medical Center ( Site 0439), Rotterdam, South Holland
  - Universitair Medisch Centrum Utrecht-Medical Oncology ( Site 0441), Utrecht
- Auckland City Hospital ( Site 0459), Auckland, New Zealand
- Oslo Universitetssykehus Ullevål ( Site 0500), Oslo, Norway
- Portugal (5):
  - Centro Hospitalar e Universitario de Coimbra ( Site 0502), Coimbra
  - Unidade Local de Saude de São José - Hospital de Santo Antonio dos Capuchos ( Site 0505), Lisbon
  - Centro Hospitalar do Porto, E.P.E. - Hospital Geral de Sto. Antonio ( Site 0504), Porto
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE ( Site 0503), Porto
  - Centro Hospitalar de Sao Joao. EPE - Hospital de Sao Joao ( Site 0501), Porto
- Puerto Rico (4):
  - Puerto Rico Medical Research Center LLC ( Site 0523), Hato Rey
  - Ad-Vance Medical Research LLC ( Site 0527), Ponce
  - VA Caribbean Healthcare System ( Site 0524), San Juan
  - FDI Clinical Research ( Site 0522), San Juan
- South Korea (10):
  - Chonnam National University Hwasun Hospital ( Site 0572), Hwasun, Jeonranamdo
  - Seoul National University Bundang Hospital ( Site 0570), Seongnam-si, Kyonggi-do
  - Pusan National University Hospital ( Site 0568), Busan, Pusan-Kwangyokshi
  - Kyungpook National University Hospital ( Site 0569), Daegu, Taegu-Kwangyokshi
  - Seoul National University Hospital ( Site 0567), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0564), Seoul
  - Asan Medical Center ( Site 0565), Seoul
  - Samsung Medical Center ( Site 0566), Seoul
  - The Catholic University of Korea St. Mary s Hospital ( Site 0571), Seoul
  - Korea University Guro Hospital ( Site 0573), Seoul
- Spain (6):
  - Hospital Universitario Puerta de Hierro ( Site 0596), Majadahonda, Madrid
  - Hospital General Universitario de Valencia ( Site 0595), Valencia, Valenciana, Comunitat
  - Hospital General Universitario Gregorio Maranon ( Site 0598), Madrid
  - Hospital Ramon y Cajal ( Site 0593), Madrid
  - Hospital Clinico San Carlos ( Site 0597), Madrid
  - Hospital Virgen del Rocio ( Site 0591), Seville
- Taiwan (8):
  - Chang Gung Medical Foundation. Kaohsiung Branch ( Site 0609), Kaohsiung City, Kaohsiung
  - Kaohsiung Medical University Hospital ( Site 0611), Kaohsiung City
  - China Medical University Hospital-Surgical Department ( Site 0610), Taichung
  - Taichung Veterans General Hospital ( Site 0613), Taichung
  - National Cheng Kung University Hospital ( Site 0608), Tainan
  - National Taiwan University Hospital ( Site 0606), Taipei
  - Taipei Veterans General Hospital-Division of Gastroenterology & Hepatology, Department of Medicine ( Site 0612), Taipei
  - Chang Gung Medical Foundation. Linkou ( Site 0607), Taoyuan District
- Thailand (3):
  - Chulalongkorn University ( Site 0627), Bangkok, Bangkok
  - Ramathibodi Hospital, Mahidol University ( Site 0628), Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital ( Site 0629), Bangkok, Bangkok
- Turkey (Türkiye) (8):
  - Hacettepe University Medical Faculty ( Site 0653), Ankara
  - Ankara City Hospital-Medical Oncology ( Site 0661), Ankara
  - Trakya University Medical Faculty Balkan Oncology Hospital ( Site 0648), Edirne
  - Bezmialem Vakf Üniversitesi-Oncology ( Site 0660), Istanbul
  - Ege University Medical Faculty Tulay Aktas Oncology Hospital ( Site 0654), Izmir
  - I.E.U. Medical Point Hastanesi ( Site 0649), Izmir
  - Konya Necmettin Erbakan University Medical Faculty ( Site 0652), Konya
  - Inonu Universitesi Medical Fakultesi ( Site 0650), Malatya
- Communal non profit enterprise Regional Clinical Oncology Center ( Site 0669), Kharkiv, Kharkivs’ka Oblast’, Ukraine
- United Kingdom (3):
  - Barts Health NHS Trust ( Site 0692), London, London, City of
  - Royal Marsden NHS Foundation Trust ( Site 0694), London, London, City of
  - Royal Marsden NHS Trust ( Site 0693), Sutton, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Kudo M, Ren Z, Guo Y, Han G, Lin H, Zheng J, Ogasawara S, Kim JH, Zhao H, Li C, Madoff DC, Ghobrial RM, Kawaoka T, Gerolami R, Ikeda M, Kumada H, El-Khoueiry AB, Vogel A, Peng X, Mody K, Dutcus C, Dubrovsky L, Siegel AB, Finn RS, Llovet JM; LEAP-012 investigators. Transarterial chemoembolisation combined with lenvatinib plus pembrolizumab versus dual placebo for unresectable, non-metastatic hepatocellular carcinoma (LEAP-012): a multicentre, randomised, double-blind, phase 3 study. Lancet. 2025 Jan 18;405(10474):203-215. doi: 10.1016/S0140-6736(24)02575-3. Epub 2025 Jan 8. PMID 39798578
- [Derived] Verset G, Borbath I, Karwal M, Verslype C, Van Vlierberghe H, Kardosh A, Zagonel V, Stal P, Sarker D, Palmer DH, Vogel A, Edeline J, Cattan S, Kudo M, Cheng AL, Ogasawara S, Daniele B, Chan SL, Knox JJ, Qin S, Siegel AB, Chisamore M, Hatogai K, Wang A, Finn RS, Zhu AX. Pembrolizumab Monotherapy for Previously Untreated Advanced Hepatocellular Carcinoma: Data from the Open-Label, Phase II KEYNOTE-224 Trial. Clin Cancer Res. 2022 Jun 13;28(12):2547-2554. doi: 10.1158/1078-0432.CCR-21-3807. PMID 35421228
- [Derived] Llovet JM, Vogel A, Madoff DC, Finn RS, Ogasawara S, Ren Z, Mody K, Li JJ, Siegel AB, Dubrovsky L, Kudo M. Randomized Phase 3 LEAP-012 Study: Transarterial Chemoembolization With or Without Lenvatinib Plus Pembrolizumab for Intermediate-Stage Hepatocellular Carcinoma Not Amenable to Curative Treatment. Cardiovasc Intervent Radiol. 2022 Apr;45(4):405-412. doi: 10.1007/s00270-021-03031-9. Epub 2022 Feb 4. PMID 35119481
- [Derived] Taylor MH, Schmidt EV, Dutcus C, Pinheiro EM, Funahashi Y, Lubiniecki G, Rasco D. The LEAP program: lenvatinib plus pembrolizumab for the treatment of advanced solid tumors. Future Oncol. 2021 Feb;17(6):637-648. doi: 10.2217/fon-2020-0937. Epub 2020 Dec 10. PMID 33300372
- [Derived] Kloeckner R, Galle PR, Bruix J. Local and Regional Therapies for Hepatocellular Carcinoma. Hepatology. 2021 Jan;73 Suppl 1:137-149. doi: 10.1002/hep.31424. Epub 2020 Nov 6. No abstract available. PMID 32557715
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26247&tenant=MT_MSD_9011